CLINICAL TRIAL: NCT03752658
Title: A Real-world Clinical Study on Effectiveness and Safety of Long-term TAF Treatment in Chronic Hepatitis B Patients in China
Brief Title: TAF Real World Study for Universal Effectiveness
Acronym: TRUE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Qin Ning, Director, Tongji Hospital
Other Study IDs: IN-US-320-4669
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, urine and whole blood will be restored in central lab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tenofovir alafenamide (TAF): Male or female HBeAg positive or negative patients (above 18 years of age) who were mono-infected with HBV, either NA treatment-naïve or treatment-experienced, but TAF naïve will be enrolled in this study, and they will be treated with TAF, alone or in combination with anti-HBV agents.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — The dose of tenofovir alafenamide (TAF) will be 25mg tablet taken orally once daily with food for 36 months, patients will be treated with TAF alone or in combination with anti-HBV agents
  Other Names: Vemlidy®

SUMMARY:
This study is a multi-center, prospective, real-world study, males and non-pregnant, non-lactating female HBeAg positive or negative patients (above 18 years of age) who were mono-infected with HBV, either NA treatment-naïve or treatment-experienced, but TAF naïve will be enrolled in this study, and they will be treated with TAF, alone or in combination with other HBV antivirals. During 36 months of treatment, efficacy and safety will be evaluated.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, real-world study, aiming to investigate the use of TAF in routine clinical management of chronic hepatitis B patients and evaluate its effectiveness and safety across a heterogeneous population in China. Approximately 500 patients will take part in this study, 10 sites will be included which distribute in China's major cities, thus each site will enroll 50 patients. Male or female HBeAg positive or negative patients (above 18 years of age) who were mono-infected with HBV, either NA treatment-naïve or treatment-experienced, but TAF naïve will be enrolled in this study, and they will be treated with TAF, alone or in combination with other HBV antivirals. During 36 months of treatment, efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Must have the ability to understand and sign a written informed consent form, consent must be obtained prior to initiation of study procedures
2. Adult males and nonpregnant, nonlactating females
3. Documented evidence of chronic HBV infection previously
4. TAF naive

Exclusion Criteria:

1. Patents who were TAF experienced
2. Women who are breastfeeding
3. Pregnant females
4. Co-infection with hepatitis A virus (HAV), hepatitis C virus (HCV), hepatitis D virus (HDV), or HIV
5. Evidence of hepatocellular carcinoma (Note: if screening alpha-fetoprotein (AFP) is < 50 ng/mL no imaging study is needed; however, if the screening AFP is > 50 ng/mL an imaging study is required)
6. Chronic liver disease of non-HBV etiology (e.g., hemochromatosis, fatty liver disease, cholangitis)
7. Current evidence of Child-Pugh Score C decompensated liver disease,or moderate to severe ascites, Grade III-IV hepatic encephalopathy
8. Abnormal hematological and biochemical parameters, including:
9. Albumin < 2.8 mg/ dL
10. International normalized ratio (INR) > 2.3 X ULN (unless stable on anticoagulant regimen)
11. Total bilirubin > 3 X ULN
12. Patient develops clinical or laboratory findings suggestive of lactic acidosis or pronounced hepatotoxicity
13. Received solid organ or bone marrow transplant, except patients who underwent liver or kidney transplantation
14. Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (e.g., basal cell skin cancer). Individuals under evaluation for possible malignancy are not eligible.
15. Individuals receiving ongoing therapy with drugs not to be used with TAF or individuals with a known hypersensitivity to study drugs, metabolites, or formulation excipients
16. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the individual unsuitable for the study or unable to comply with dosing requirements
17. Use of investigational agents within 3 months of screening, unless allowed by the sponsor
18. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening
19. Current alcohol or substance abuse judged by the investigator to potentially interfere with compliance
20. Inability or unwillingness to provide informed consent or abide by the requirements of the study
21. In addition to the above exclusion criteria, patients who meet any of the contraindications for TAF

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and non-pregnant, non-lactating female patients with HBsAg positive > 6 months above 18 years of age; Documented evidence of chronic HBV infection previously; HBV mono-infected HBeAg positive or negative; NA treatment-naive and treatment-experienced; TAF naive; Agree to participate in the study and sign the patient informed consent.
  Subjects coinfected with HCV, hepatitis D virus (HDV), human immunodeficiency virus (HIV) or who have received TAF or who haveChild-Pugh C decompensated liver disease or HCC will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
proportion of participants with HBV DNA < 20 IU/mL | 36 months
  proportion of participants with HBV DNA < 20 IU/mL as measured by the COBAS TaqMan HBV Test (Roche Molecular Diagnostics, Pleasanton, CA, USA), with taken at 36 months

SECONDARY OUTCOMES:
The proportion of patients with HBV DNA < 20 IU/mL | 12 months
  The proportion of patients with HBV DNA < 20 IU/mL at 12 months
The proportion of patients with HBV DNA <300 copies/mL | 12 months
  The proportion of patients with HBV DNA <300 copies/mL at 12 months
The proportion of patients with HBV DNA < 20 IU/mL | 24 months
  The proportion of patients with HBV DNA < 20 IU/mL at 24 months
The proportion of patients with HBV DNA <300 copies/mL IU/mL | 24 months
  The proportion of patients with HBV DNA <300 copies/mL at 24 months
The proportion of patients with HBV DNA <300 copies/mL IU/mL | 36 months
  The proportion of patients with HBV DNA <300 copies/mL at 36 months
Proportion of participants with Hepatitis B e Antigen (HBeAg) Loss | 36 months
  Proportion of participants with Hepatitis B e Antigen (HBeAg) Loss at 36 months
Proportion of participants with seroconversion to Anti-Hepatitis B e-Antigen (Anti-HBe) | 36 months
  Proportion of participants with seroconversion to Anti-Hepatitis B e-Antigen (Anti-HBe) at 36 months
Proportion of participants with Normal Alanine Aminotransferase (ALT) | 36 months
  Proportion of participants with Normal Alanine Aminotransferase (ALT) at 36 months
Change from baseline in fibrosis as assessed by Fibroscan® | 36 months
  Change from baseline in fibrosis as assessed by Fibroscan® at 36 months
Percent Change from baseline in Bone Mineral Density (BMD) | 36 months
  Percent Change from baseline in Bone Mineral Density (BMD) at 36 months
Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) | 36 months
  Change from baseline in Estimated Glomerular Filtration Rate by the Cockcroft-Gault Formula (eGFR-CG) at 36 months
the rate of mother-to-child transmission of HBV | at postpartum 6 months
  For unplanned pregnant subjects, if not withdrawn, mother-to-child transmission (MTCT) rate

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, MD., Ph.D., Study Chair — Department and Institute of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (7):
- China (7):
  - Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Shulan(Hangzhou) hospitai, Hangzhou
  - First Affiliated Hospital of Nanchang University, Nanchang
  - Shanghai public health clinic, Shanghai
  - General Hospital of The Yangtze River Shipping, Wuhan
  - The Seventh Hospital of Wuhan, Wuhan
  - Xiangya Hospital of Central South University, Xiangya